CLINICAL TRIAL: NCT05950321
Title: Comparison of Fluoroscopy-guided Cervical Paramedian Interlaminar Epidural Block Versus Ultrasound-guided Selective Nerve Root Pulsed Radiofrequency for the Management of Chronic Lower Cervical Radicular Pain
Brief Title: Paramedian CESI vs Selective Nerve Root PRF for Lower Cervical Radicular Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Supervisor Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Paramedian cesi vs root prf
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Neck Pain; Cervical Radiculopathy
Keywords: Pulsed Radiofrequency Treatment; Fluoroscopy; Steroids
MeSH Terms: conditions — Neck Pain; Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cervical epidural group (Active Comparator): Paramedian cervical epidural injection for cervical radiculopathy
  Interventions: Procedure: Paramedian cervical epidural steroid injection
- Radiofrequency group (Active Comparator): Pulsed radiofrequency applied to nerve roots for cervical radiculopathy
  Interventions: Procedure: Selective nerve root pulsed radiofrequency

INTERVENTIONS:
Procedure: Paramedian cervical epidural steroid injection — For paramedian cervical epidural steroid injection, the cervical 7 (C7) - thoracic 1 (T1) interval is determined by taking an appropriate angle with C-arm fluoroscopy to determine the interlaminar space from the posterior cervical region. The epidural space is recognized by the negative pressure reflected on the resistance syringe.
  Arms: Cervical epidural group
Procedure: Selective nerve root pulsed radiofrequency — For selective nerve root PRF, an 8-12 Hz linear ultrasound probe is first placed posterolateral to the neck. The level of the cervical nerve roots is determined according to the morphology of the anterior and posterior vertebral tubercles. The corresponding nerve root is visualized hypoechoically between the tubercles. The radiofrequency cannula is inserted in the same plane as the ultrasound probe (in plane) and the relevant nerve root is approached. Pulsed radiofrequency current, which has therapeutic properties in chronic pain, is applied to the relevant nerve root for 240 seconds.
  Arms: Radiofrequency group

SUMMARY:
This study aims to compare the efficacy of ultrasound-guided selective cervical nerve root pulsed radiofrequency (PRF) versus fluoroscopy-guided paramedian cervical epidural steroid administration (CESI) for the treatment of lower cervical radicular pain refractory to conservative treatments. For this evaluation, a numerical rating (NRS), neck disability index (NDI), and Leeds Assessment Of Neuropathic Symptoms And Signs (LANSS) scale will be used before and after both interventions.

DETAILED DESCRIPTION:
Chronic cervical radicular pain is a common condition that affects the quality of life of many patients and is caused by compression or irritation of the cervical nerve roots. Treatment options for this condition include conservative methods such as medications and physical therapy, as well as interventions such as surgery or injections.

Two commonly used injections for chronic cervical radicular pain are ultrasound-guided selective nerve root PRF and fluoroscopy-guided paramedian CESI. PRF involves the application of pulsed radiofrequency energy (intermittent current, tissue temperature not exceeding 42 °C) to the cervical nerve root under ultrasound guidance. PRF is a non-destructive technique that modulates the activity of nerve fibers without causing thermal damage. CESI involves injecting local anesthetic and steroids into the epidural space between the laminae of the vertebrae under fluoroscopic guidance. The aim of both techniques is to reduce inflammation and pain transmission from the affected nerve root. The efficacy of both CESI and selective nerve root PRF has been demonstrated in clinical trials.

The primary aim of the investigators in this study is to compare the efficacy of these two treatments. A total of at least 60 patients, 30 patients in each group, will be enrolled for comparison. NRS, NDI, and LANSS scores before, 3 months, and 6 months after treatment will be compared both within and between groups. The secondary aim is to reveal the side effects and adverse events in these two treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Severe unilateral radicular pain due to cervical disc herniation (pain with a severity of 6 or more on a numeric rating scale of 0-10)
* Continued pain for more than 3 months
* Demonstration of herniated disc compression of the lower cervical spinal nerve roots on magnetic resonance imaging
* Failure in pain management with conservative methods such as analgesics and physical therapy

Exclusion Criteria:

* Pain radiating to both arms, hands or neck pain in the foreground
* Spinal stenosis or spondylolisthesis (only those with radicular pain due to disc herniation will be included)
* Cognitive impairment
* Hepatic or renal insufficiency
* Severe psychiatric illness
* Local or systemic infection
* Coagulopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) | Change from baseline to 3rd and 6th month after treatment
  NRS is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain)

SECONDARY OUTCOMES:
The Neck Disability Index (NDI) | Change from baseline to 3rd and 6th month after treatment
  The Neck Disability Index (NDI) is a widely used questionnaire designed to assess the impact of neck pain on a person's daily functioning and quality of life. It consists of ten questions covering topics such as pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each question has six possible responses, which are assigned a numerical value. By summing up the scores, the NDI provides a measure of the patient's neck disability ranging from 0% (no disability) to 100% (maximum disability).
Leeds Assessment Of Neuropathic Symptoms And Signs (LANSS) | Change from baseline to 3rd and 6th month after treatment
  The Leeds assessment of neuropathic symptoms and signs (LANSS) Pain Scale is based on analysis of sensory description and bedside examination of sensory dysfunction, and provides immediate information in clinical settings. It was developed in two populations of chronic pain patients.

CONTACTS AND LOCATIONS:
Overall Officials: Gevher Rabia Genc Perdecioğlu, Study Chair — Diskapi TRH
Locations (1):
- Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)